CLINICAL TRIAL: NCT07349173
Title: Study of the Representation of Action Peripersonal Space in Participants With Unilateral Segmental Exclusion of the Upper Limb Compared to Asymptomatic Subjects
Brief Title: Peripersonal Space Representation in Upper Limb Segmental Exclusion
Status: Not yet recruiting | Type: Observational
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Responsible Party: Sponsor
Other Study IDs: IRR-CLP-2023-3; 2025-A02189-40 (Other: ID-RCB)
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Segmental Exclusion Syndrome; Complex Regional Pain Syndrome (CRPS); Upper Limb Neglect (Peripheral)
Keywords: Peripersonal Space; Virtual Reality; Body Schema; Reachability Judgment
MeSH Terms: conditions — Complex Regional Pain Syndromes; Personal Space

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Exclusion: Patients presenting with unilateral segmental exclusion of the upper limb or part of the hand evolving for more than 3 months.
  Interventions: Behavioral: Reachability Judgment Task in VR.
- Healthy Controls: symptomatic volunteers with no history of upper limb impairment with sequelae.
  Interventions: Behavioral: Reachability Judgment Task in VR.

INTERVENTIONS:
Behavioral: Reachability Judgment Task in VR. — Participants wear an Oculus Quest 2 VR headset. They first perform a motor task to measure Real Reachable Distance (DMA-r). Then, they perform a perceptual task where they must judge, without moving, if a virtual object is reachable (DMA-p). The test evaluates different spatial planes (front, 45° right, 45° left) and heights (shoulder, navel).

SUMMARY:
This study aims to evaluate the representation of action peripersonal space (PPS) in subjects suffering from unilateral segmental exclusion syndrome of the upper limb compared to healthy control subjects. Segmental exclusion is defined by non-use or under-use of a limb segment without central nervous system damage. The study hypothesizes that this syndrome leads to a modification (shrinkage) of the PPS representation. Participants will perform reachability judgments in a Virtual Reality (VR) environment.

DETAILED DESCRIPTION:
Segmental exclusion syndrome often occurs after limb trauma and manifests as a neglect-like behavior of peripheral origin, sometimes associated with Complex Regional Pain Syndrome (CRPS). The study explores whether the lack of limb use affects the representation of peripersonal space (PPS)-the space immediately surrounding the body where interactions with objects occur.

The study is monocentric, observational, with a matched control group. Participants will undergo:

Clinical assessment (questionnaires on pain, anxiety, body perception, and kinesiophobia).

A Virtual Reality (VR) test (approx. 40 minutes). In VR, participants will judge whether a cylinder presented at different distances and angles is reachable without moving (Perceived Reachable Distance - DMA-p). This will be compared to their Real Reachable Distance (DMA-r).

The goal is to measure the error of judgment to assess PPS representation and check for correlations with body schema disturbances or functional impairment

ELIGIBILITY:
Inclusion Criteria (patients):

* Age ≥ 18 years.
* Presenting unilateral exclusion symptom of the upper limb or part of the hand evolving for > 3 months.
* No contraindication to force work in daily activities.
* For patients with finger exclusion: at least 2 perturbed items related to exclusion on tests 3 and 4 of the "Bilan 400 points".
* Affiliated to a social security scheme.
* Able to understand simple orders.

Inclusion Criteria (Controls):

* Age ≥ 18 years.
* No history of upper limb impairment with sequelae.

Exclusion Criteria (All):

* Visual impairments.
* Central neurological pathology.
* Unstabilized psychiatric pathology.
* Communication or comprehension difficulties.
* Under legal protection or unable to consent.
* Pregnant or breastfeeding women.
* Cervical pathology contraindicating VR headset use.
* Epilepsy.
* Upper limb pathology unrelated to exclusion.
* Inability to stand for 40 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: he study population consists of two groups recruited at the Institut Régional de Réadaptation (Centre Louis Pierquin, UGECAM Nord-Est) in Nancy, France.
  Patients with Exclusion: Participants are selected from patients receiving routine care (full hospitalization or day hospital) at the center. They are identified based on a functional assessment ("Bilan 400 points") showing specific impairments related to unilateral upper limb exclusion evolving for more than 3 months.
  Healthy Controls: Asymptomatic volunteers are recruited through the social or family network of the investigators and current participants, as well as via posters displayed in the UGECAM centers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Judgment Error of Reachability | Day 1 (During the 40-minute VR assessment)
  Difference between Perceived and Real Reachable Distance. Calculated as the normalized difference between the Perceived Maximum Reachable Distance (DMA-p) and the Real Maximum Reachable Distance (DMA-r). Formula: ((DMA-p - DMA-r) / DMA-r) * 100. This assesses the overestimation or underestimation of the peripersonal space.

SECONDARY OUTCOMES:
Body Perception Disturbance Score | Day 1 (Before VR task)
  Assessed using the Bath CRPS Body Perception Disturbance Scale (French version). Scores range from 0 to 57, with higher scores indicating greater disturbance.
Functional Impairment Score (400-Point Hand Assessment) | Day 1
  Evaluation of functional hand use (score and number of perturbed items).
Anxiety and Depression Score (HAD) | Day 1
  Hospital Anxiety and Depression Scale. Scores range from 0 to 21 for each dimension (Anxiety and Depression).
Kinesiophobia Score (Tampa Scale) | Day 1
  Tampa Scale for Kinesiophobia (TSK). Assesses fear of movement. Scores range to 68; >40 indicates significant kinesiophobia.
Pain Catastrophizing Score (PCS) | Day 1
  Pain Catastrophizing Scale. Scores range from 0 to 52.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation (IRR), Centre Louis Pierquin., Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided